CLINICAL TRIAL: NCT02380755
Title: Clomiphene Citrate for the Treatment of Obesity Related Male Hypogonadism: Metabolic and Cardiovascular Effects.
Brief Title: Clomiphene Citrate for the Treatment of Obesity Related Male Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Cintia Cercato, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 385.615; 2013/16781-1 (Other: FAPESP)
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Hypoandrogenism
Keywords: Flow-mediated dilatation; Clomiphene citrate; sICAM-1; sVCAM-1; sE- Selectin; Endothelial function; Cardiovascular risk; Endocrine System Diseases; Selective Estrogen Receptor Modulators; Estrogen Receptor Modulators; Infertility, Male; Endothelial Progenitor Cells; Obesity; Testosterone
MeSH Terms: conditions — Obesity; Endocrine System Diseases; Infertility, Male | interventions — Clomiphene

STUDY DESIGN:
Intervention Model Description: 78 patients were randomized (1:1) to receive Clomiphene Citrate (CC) 50 mg during 12 weeks or placebo (PLB). MAIN OUTCOME MEASURES: flow-mediated dilatation of the brachial artery (FMDAB), circulating levels of sICAM-1, sVCAM-1, E-selectin and progenitor endothelial cells. Secondary endpoints: Body mass index (BMI), abdominal circumference (AC), glycaemia, total cholesterol, fractions and triglycerides, HOMA-IR index, bioelectrical impedance parameters, Adam questionnaire and hormonal parameters (total testosterone levels, SHBG, LH, FSH and Estradiol).
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomized, double blinded, placebo-controlled, parallel group, single-center study
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): One pill every other day during 12 weeks
  Interventions: Drug: Placebo
- Clomiphene Citrate (Active Comparator): Clomiphene citrate 50 mg orally daily (Serophene) during 12 weeks
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Clomiphene Citrate — 50 mg orally daily during 12 weeks
  Other Names: Serophene
  Arms: Clomiphene Citrate
Drug: Placebo — 1 pill orally daily during 12 weeks
  Other Names: Control
  Arms: Placebo

SUMMARY:
Hypogonadism is a clinical condition that can be associated with obesity in man. Controversy exists regarding if its a condition that needs to be treated. The standard Testosterone Therapy is associated with increase in cardiovascular risks, according to some studies, and leads to infertility. The use of Clomiphene Citrate in this sub population of obese man as an alternative treatment option is not well studied. The aim of this protocol is to evaluate the cardiovascular risks, metabolic and hormonal parameters in a double blinded randomized placebo trial.

DETAILED DESCRIPTION:
Hypogonadism (low testosterone level) in obese man is a clinical condition which treatment is controversial. Most of this controversy remains regarding the association between cardiovascular risk elevation and Testosterone replacement therapy in some studies.

This protocol is a double blinded randomized placebo trial and 2 groups will be followed. The primary end-point of this research is the correlation between the serum testosterone and flow-mediated dilatation of the brachial artery (FMDAB), circulating levels of sICAM-1, sVCAM-1, E-selectin and progenitor endothelial cells.

The secondary end-points include:

(1) the evaluation of metabolic parameters: weight, abdominal circumference, glycaemia, total cholesterol, fractions and triglycerides, homeostasis model assessment index (HOMA) and bioelectrical impedance parameters; and (2) hormonal parameters: total testosterone levels, sex hormone-binding globulin (SHBG), Luteinizing Hormone (LH) , Follicle stimulating hormone (FSH) and Estradiol.

ELIGIBILITY:
Inclusion Criteria:

* ADAM questionnaire positive for 3 or more questions
* Total serum Testosterone lower than 300 ng/dL in two different occasions, within a 1-week minimum interval. This blood sample must be collected between 8 and 11 a.m.
* Low or Inappropriate normal serum Luteinizing hormone (LH) level
* ATP III Metabolic Syndrome Criteria
* Obesity - BMI over 30 kg/m2

Exclusion Criteria:

* Systemic illness, such Rheumatoid Arthritis, Cushing disease, liver insufficiency or renal insufficiency. -Use of certain medications (opiates, high-dose glucocorticoid therapy, methadone)
* Eating disorders
* Testicular volume below 4 mL
* Use of recreational drugs
* Excessive exercise practice
* Men in treatment for prostatic cancer
* Hyperprolactinaemia
* Hemochromatosis
* History of headache
* Systolic blood pressure lower than 100 mmHg
* Previous adverse reactions to nitrate compounds
* Diabetes over 10 years of diagnosis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | baseline up to 12 weeks
  1. Flow-mediated dilatation of the brachial artery (FMDAB): Brachial artery FMD is calculated as the percentage increase in brachial artery diameter with hyperemia induced relative to the resting brachial artery diameter. Percentage of brachial artery diameter is measured as FMD diameter/basal diameter.
  2. Icam, vcam and selectin
  3. Endothelial progenitor cels
Total Testosterone | baseline up to 12 weeks
  electrochemical luminescence analysis in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Cintia Cercato, MD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da USP; Elaine Maria F Costa, Prof, PhD, Principal Investigator — Faculdade de Medicina da USP
Locations (1):
- Prédio dos ambulatórios HCFMUSP - PAMB, São Paulo, Brazil